CLINICAL TRIAL: NCT01338519
Title: Database Study on Patients With PCOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Other Study IDs: PCOSDatabaseOdense
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 1997-01

CONDITIONS: Hirsutism; PCOS
MeSH Terms: conditions — Hirsutism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCOS and hirsutism

SUMMARY:
All newly referred patients with PCOS and hirsutism are listed in a database.

DETAILED DESCRIPTION:
All premenopausal women referred to the outpatient clinic at the Department of Endocrinology from 1997 and onward with the referral diagnoses hirsutism and/or PCOS are included in a clinical database. The patients should fulfill the Rotterdam criteria for PCOS or have clinical/biochemical hyperandrogenemia.

Routine evaluation include medical history, clinical examination, transvaginal ultrasound (US), and fasting blood samples. Cycle history is recorded in all patients using a standard scheme prepared for hirsute patients. Blood tests include androgens, LH, FSH, prolactin, and lipid profile.

OGTT and ACTH are performed in high risk patients

ELIGIBILITY:
Inclusion Criteria:

* premenopausal
* hirsutism or PCOS

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Premenopausal women referred with hirsutism or PCOS to Odense University hospital
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1997-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, MD, PhD, Principal Investigator — Odense Univeristy Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark